CLINICAL TRIAL: NCT04601272
Title: Evaluating the Performance of the Shared Decision Making Process Scale in Patients Making Cancer Screening Decisions
Brief Title: Evaluating the Shared Decision Making Process Scale in Cancer Screening Decisions
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Sepucha, Director, Health Decision Sciences Center, Massachusetts General Hospital
Other Study IDs: 2005P002282
Record Dates: First submitted 2020-09-29; First posted 2020-10-23 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer Screening; Colon Cancer Screening; Prostate Cancer Screening
Keywords: decision making; decision aids; decision quality instruments; shared decision making; cancer screening
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast Cancer Screening: Women between the ages of 35-55 when they received a decision aid for breast cancer screening with no prior diagnosis of breast cancer. These people will see items only pertaining to breast cancer screening.
  Interventions: Behavioral: Decision aid
- Colon Cancer Screening: Men and women between the ages of 45-75 when they received a decision aid for colon cancer screening with no prior diagnosis of colon cancer. These people will see items only pertaining to colon cancer screening.
  Interventions: Behavioral: Decision aid
- Prostate Cancer Screening: Men between the ages of 45-74 when they received a decision aid for prostate cancer screening with no prior diagnosis of prostate cancer. These people will see items only pertaining to prostate cancer screening.
  Interventions: Behavioral: Decision aid

INTERVENTIONS:
Behavioral: Decision aid — Healthwise patient decision aids for breast, prostate, colon and lung cancer screening provide information on the pros and cons of cancer screening and guidance in process of selecting a choice.

SUMMARY:
The purpose of this retrospective observational study is to evaluate the performance of the Shared Decision Making Process scale in a sample of patients who have received a decision aid about the decision to screen or not screen for breast cancer, colon cancer, prostate cancer, or lung cancer.

DETAILED DESCRIPTION:
This is a retrospective observational study that will examine the performance of the Shared Decision Making Process in a sample of patients who made a decision about cancer screening in the last 2 years. Patients from 4 hospitals who have received a patient decision aid for breast, colon, prostate, or lung cancer screening will be screened for eligibility. A random sample of eligible patients will be sent a one-time survey. The survey asks patients about their experiences talking with healthcare providers about the specific cancer screening decision. The survey includes the Shared Decision Making Process scale, knowledge, preferences, decisional conflict and decision regret. The study will obtain 400 completed surveys, or 100 for each cancer topic.

The sample consists of patients who received a decision aid for cancer screening within the last two years and meet specific qualifications.

All analyses will be conducted separately for each group, and results may be pooled. First, study staff examine the descriptives for the Shared Decision Making Process items. Study staff will also test several hypotheses to examine performance of the scores such as whether higher shared decision making process scores are associated with less decisional conflict and less regret.

ELIGIBILITY:
Inclusion Criteria:

Breast Cancer group

* Female sex
* Between ages of 35-55
* No previous diagnosis of breast cancer

Colon Cancer Group

* Between ages of 45-75
* No previous diagnosis of colon cancer

Prostate Cancer Group

* Male sex
* Between ages of 45-74
* No previous diagnosis of prostate cancer

Lung Cancer Group

* Between ages of 50-80
* No previous diagnosis of lung cancer

Exclusion Criteria:

Breast Cancer group

* Unable to confirm primary language is English
* History of breast cancer
* Severe cognitive impairment who cannot consent for themselves

Colon Cancer Group

* Unable to confirm primary language is English
* History of colon cancer
* Severe cognitive impairment who cannot consent for themselves

Prostate Cancer Group

* Unable to confirm primary language is English
* History of prostate cancer
* Severe cognitive impairment who cannot consent for themselves

Lung Cancer Group

* Unable to confirm primary language is English
* History of lung cancer
* Severe cognitive impairment who cannot consent for themselves

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who received a cancer screening decision aid in the last 2 years while receiving care at 4 hospitals within a major healthcare network.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen R Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will create a complete, cleaned, de-identified copy of the final data set for each cancer screening topic.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be made available to outside investigators starting 6 months after publication.
Access Criteria: Information about the data sets will be on the Health Decision Sciences Center website and in publications of the data. Dr. Sepucha will share a de-identified data set with outside investigators at no cost, according to approved Massachusetts General Hospital (MGH)/ Partners policies for datasharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board (IRB) requirements are met before using the data,that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were Mass General Brigham patients who were ordered a Decision Aid between July 2018 and December 2020 for one of the 3 cancer screening topics: breast, colon, or prostate.
Pre-assignment Details: Eligible patients were English speaking and fell within the appropriate age range for considering cancer screening for the clinical topic. Colon cancer group were patients between 45 and 75 years old; breast cancer group were women between 35 and 55 years old; prostate cancer group were men between 45 and 74 years old.
Period: Overall Study
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Started | 73 | 89 | 78
Completed | 71 | 86 | 76
Not Completed | 2 | 3 | 2
Not completed — did not have sufficient information to calculate the SDM Process score (primary outcome) | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Participants who received a decision aid for breast/colon/prostate cancer within the last 2 years. Participants provided enough information to calculate the shared decision making process score (primary outcome of interest)
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening | Total
Number analyzed (Participants) | 71 | 86 | 76 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (4) | 60 (9) | 59 (8) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 60 | 76 | 207
  Male | 0 | 26 | 0 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 8
  Not Hispanic or Latino | 67 | 56 | 71 | 194
  Unknown or Not Reported | 1 | 27 | 3 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 5 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 2 | 8
  White | 48 | 73 | 66 | 187
  More than one race | 2 | 3 | 0 | 5
  Unknown or Not Reported | 3 | 4 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 71 | 86 | 76 | 334

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making Process Measure
Description: The Shared Decision Making Process is a short patient-reported survey that measures the amount of shared decision making that occurs in an interaction. Scores range from 0-4 where higher values indicate a better shared decision making process outcome.
Time Frame: Baseline survey
Population: participants who provided enough information to calculate a shared decision making process score (primary outcome of interest). 233/233 patients provided an answer to this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 71 | 86 | 76
score on a scale | 1.05 (1.07) | 1.20 (1.10) | 2.10 (0.90)

2. Secondary Outcome: The 9-item Shared Decision Making Questionnaire
Description: The Shared Decision Making Questionnaire measure measures the amount of shared decision making that occurs in an interaction. Scores range from 0-100 where higher values indicate a better shared decision making process occurred.
Time Frame: Baseline survey
Population: participants who answered at least 2 out of 9 of the 9-item shared decision making questionnaire. Only 223/233 participants provided sufficient information to calculate a SDMQ9 score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 69 | 82 | 72
score on a scale | 50.5 (25.6) | 56.8 (27.9) | 63.8 (22.9)

3. Secondary Outcome: Decisional Conflict Tool (SURE)
Description: Measures decisional conflict, consists of 4 yes/no items. Scores range 0-4 where 0 indicates extremely high decisional conflict, 4 indicates no decisional conflict. The number who get score of 4 is reported indicating no decisional conflict.
Time Frame: Baseline survey
Population: participants who answered all 4 items of the decisional conflict scale. Only 217/233 provided sufficient information to calculate a SURE score.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 69 | 78 | 70
percentage of participants | 49 | 51 | 67

4. Secondary Outcome: Single-Item Measure of Decision Regret
Description: Single item asking "If you knew then what you know now, do you think you would make the same decision about [breast cancer screening/colon cancer screening/ prostate cancer screening/lung cancer screening]?" where the last part varies by group.
  Response options are:
  Definitely yes, Probably yes, Probably No, Definitely No
Time Frame: Baseline survey
Population: Participants who answered the single-item regret question. Only 220/233 participants provided sufficient information to calculate regret.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 65 | 84 | 71
Participants
  Definitely yes | 33 | 44 | 33
  Probably yes | 27 | 32 | 32
  Probably no | 3 | 6 | 6
  Definitely no | 2 | 2 | 0

5. Secondary Outcome: Treatment Choice
Description: Single item asking patient "What did you want to do" in regard to (depending on the group) colon cancer screening/ breast cancer screening/ prostate cancer screening/ lung cancer screening.
Time Frame: Baseline survey
Population: Participants who answered the question asking their treatment preference. Only 231/233 provided sufficient information for this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 71 | 86 | 74
Participants
  Start mammograms in 40s | 39 | NA — response option only administered to breast cancer screening group | NA — response option only administered to breast cancer screening group
  Wait until 50 | 8 | NA — response option only administered to breast cancer screening group | NA — response option only administered to breast cancer screening group
  Have a colonoscopy | NA — response option only administered to colon cancer screening group | 45 | NA — response option only administered to colon cancer screening group
  Do a stool-based test | NA — response option only administered to colon cancer screening group | 24 | NA — response option only administered to colon cancer screening group
  No screening | NA — response option only administered to colon cancer screening group | 1 | NA — response option only administered to colon cancer screening group
  Have a PSA test | NA — response option only administered to prostate cancer screening group | NA — response option only administered to prostate cancer screening group | 42
  Not have a PSA test | NA — response option only administered to prostate cancer screening group | NA — response option only administered to prostate cancer screening group | 20
  Do something else | 10 | 8 | 1
  Unsure | 14 | 8 | 11

6. Secondary Outcome: Adapted Controlled Preference Scale
Description: Single item asking the participants who made the ultimate decision. The categorical response options are:
  1. the patient made the decision
  2. the provider made the decision
  3. both patient and provider made the decision together.
Time Frame: Baseline survey
Population: participants who answered the adapted controlled preference question. Only 220/233 participants provided sufficient information to calculate preference.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 66 | 82 | 72
Participants
  Mainly my decision | 33 | 33 | 45
  Mainly the healthcare providers decision | 10 | 19 | 5
  We made the decision together | 23 | 30 | 22

7. Secondary Outcome: Knowledge
Description: Multiple choice knowledge items specific for each topic will be combined to a total knowledge score (0-100) with higher scores indicating higher knowledge. These items are part of the knowledge subscale in the published Decision Quality Instruments.
Time Frame: Baseline survey
Population: participants who completed at least 60% of the knowledge questions for their respective cancer screening group. Only 225/233 participants provided sufficient information to calculate a knowledge score.
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 71 | 84 | 70
percentage of correct answers | 43 (21) | 58 (19) | 62 (24)

ADVERSE EVENTS:
Time Frame: The surveys were reviewed within 2 weeks as they came in for evidence of adverse events.
Arm/Group | Breast Cancer Screening | Colon Cancer Screening | Prostate Cancer Screening
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/86 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/86 | 0/76
Other Adverse Events (participants affected / at risk) | 0/71 | 0/86 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04601272/Prot_SAP_000.pdf